CLINICAL TRIAL: NCT04786769
Title: A Randomized Clinical Trial of Intravenous Iron Supplementation in TAVI and SAVR Patients With Iron Deficiency
Brief Title: Iron Supplementation in TAVI and SAVR Patients With Iron Deficiency
Acronym: INERTIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Santa Cruz, Portugal (Other)
Responsible Party: Principal Investigator, Afonso Félix de Oliveira, Principal Investigator, Hospital de Santa Cruz, Portugal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNICARV-1
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Aortic Stenosis; Iron-deficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Two-arm trial of intravenous iron supplementation vs placebo, randomized 1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron supplementation (Experimental): Intravenous ferric carboxymaltose will be administered according to weight and hemoglobin values at randomization as follows:
  2-4 weeks before valve intervention On the day of admission to valve intervention (if determined by dose calculation, otherwise placebo) 12 weeks after valve intervention (if iron deficiency persists, otherwise placebo)
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Intravenous 0.9% NaCl (placebo) will be administered as follows:
  2-4 weeks before valve intervention On the day of admission to valve intervention 12 weeks after valve intervention
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous ferric carboxymaltose according to baseline weight and hemoglobin

SUMMARY:
The INERTIA trial is a multicenter double-blinded randomized trial of intravenous iron supplementation in patients with severe aortic stenosis and iron deficiency undergoing TAVI or SAVR. The primary endpoint is the time to HF hospital admission or cardiovascular death. Secondary endpoints will assess quality of life indicators and functional capacity at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis
* Enrolled for TAVI or SAVR procedures
* Documented iron deficiency with either: Ferritin <100ug/L or Ferritin between 100-299ug/L and Transferrin Saturation < 20%.

Exclusion Criteria:

* Use of packed red blood cells or whole blood in the past 3 months;
* Use of erythropoietin-stimulating agent or IV iron in the past 3 months;
* Use of oral or IV iron (>100mg/day) in the past 3 months;
* Haemoglobin (Hb) levels > 15g/dL or < 8g/dL;
* Active cancer;
* Infection requiring antibiotic treatment at the time of first scheduled dose;
* Any known contraindication to study intervention

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with heart failure hospital admission or cardiovascular death | up to 52 weeks
  Analyzed as time-to-event

SECONDARY OUTCOMES:
Total number of allogeneic RBC units received | 30 days post-TAVI or SAVR
Walking distance | 6 months post-TAVI or SAVR
  6 minute walking test
Kansas City Cardiomyopathy Questionnaire | 6 months post-TAVI or SAVR
  Heart failure symptoms assessment. 0-100 scale, higher scores reflect better health status.
Patient Global Assessment | 6 months post-TAVI or SAVR
  Patient reported outcome on the impact of the disease in daily live
EQ-5D-5L | 6 months post-TAVI or SAVR
  Quality of life assessment in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Afonso Félix-Oliveira, MSc, Principal Investigator — Hospital de Santa Cruz, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroll JD, Mack MJ, Vemulapalli S, Herrmann HC, Gleason TG, Hanzel G, Deeb GM, Thourani VH, Cohen DJ, Desai N, Kirtane AJ, Fitzgerald S, Michaels J, Krohn C, Masoudi FA, Brindis RG, Bavaria JE. STS-ACC TVT Registry of Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2020 Nov 24;76(21):2492-2516. doi: 10.1016/j.jacc.2020.09.595. PMID 33213729
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Vemulapalli S, Dai D, Hammill BG, Baron SJ, Cohen DJ, Mack MJ, Holmes DR Jr. Hospital Resource Utilization Before and After Transcatheter Aortic Valve Replacement: The STS/ACC TVT Registry. J Am Coll Cardiol. 2019 Mar 19;73(10):1135-1146. doi: 10.1016/j.jacc.2018.12.049. PMID 30871697
- [Background] Myles PS, Richards T, Klein A. Preoperative intravenous iron for cardiac surgery. Lancet. 2020 Dec 12;396(10266):1883-1884. doi: 10.1016/S0140-6736(20)32406-5. No abstract available. PMID 33308468
- [Background] Abdul-Jawad Altisent O, Puri R, Regueiro A, Chamandi C, Rodriguez-Gabella T, Del Trigo M, Campelo-Parada F, Couture T, Marsal JR, Cote M, Paradis JM, DeLarochelliere R, Doyle D, Mohammadi S, Dumont E, Rodes-Cabau J. Predictors and Association With Clinical Outcomes of the Changes in Exercise Capacity After Transcatheter Aortic Valve Replacement. Circulation. 2017 Aug 15;136(7):632-643. doi: 10.1161/CIRCULATIONAHA.116.026349. Epub 2017 Jun 6. PMID 28588077
- [Background] Zimarino M, Barbanti M, Dangas GD, Testa L, Capodanno D, Stefanini GG, Radico F, Marchioni M, Amat-Santos I, Piva T, Saia F, Reimers B, De Innocentiis C, Picchi A, Toro A, Rodriguez-Gabella T, Nicolini E, Moretti C, Gallina S, Maddestra N, Bedogni F, Tamburino C. Early Adverse Impact of Transfusion After Transcatheter Aortic Valve Replacement: A Propensity-Matched Comparison From the TRITAVI Registry. Circ Cardiovasc Interv. 2020 Dec;13(12):e009026. doi: 10.1161/CIRCINTERVENTIONS.120.009026. Epub 2020 Dec 4. PMID 33272037
- [Background] Costa F, Cohen MG. Transfusion and Mortality After Transcatheter Aortic Valve Replacement: Association or Causation? Circ Cardiovasc Interv. 2020 Dec;13(12):e010225. doi: 10.1161/CIRCINTERVENTIONS.120.010225. Epub 2020 Dec 4. No abstract available. PMID 33272032
- [Background] Nuis RJ, Rodes-Cabau J, Sinning JM, van Garsse L, Kefer J, Bosmans J, Dager AE, van Mieghem N, Urena M, Nickenig G, Werner N, Maessen J, Astarci P, Perez S, Benitez LM, Dumont E, van Domburg RT, de Jaegere PP. Blood transfusion and the risk of acute kidney injury after transcatheter aortic valve implantation. Circ Cardiovasc Interv. 2012 Oct;5(5):680-8. doi: 10.1161/CIRCINTERVENTIONS.112.971291. Epub 2012 Oct 9. PMID 23048055
- [Background] Klein AA, Chau M, Yeates JA, Collier T, Evans C, Agarwal S, Richards T; UK Cardiac and Vascular Surgery Interventional Anaemia Response (CAVIAR) study team. Preoperative intravenous iron before cardiac surgery: a prospective multicentre feasibility study. Br J Anaesth. 2020 Mar;124(3):243-250. doi: 10.1016/j.bja.2019.11.023. Epub 2020 Jan 3. PMID 31902590
- [Background] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Background] Ponikowski P, van Veldhuisen DJ, Comin-Colet J, Ertl G, Komajda M, Mareev V, McDonagh T, Parkhomenko A, Tavazzi L, Levesque V, Mori C, Roubert B, Filippatos G, Ruschitzka F, Anker SD; CONFIRM-HF Investigators. Beneficial effects of long-term intravenous iron therapy with ferric carboxymaltose in patients with symptomatic heart failure and iron deficiencydagger. Eur Heart J. 2015 Mar 14;36(11):657-68. doi: 10.1093/eurheartj/ehu385. Epub 2014 Aug 31. PMID 25176939
- [Background] Jankowska EA, Tkaczyszyn M, Suchocki T, Drozd M, von Haehling S, Doehner W, Banasiak W, Filippatos G, Anker SD, Ponikowski P. Effects of intravenous iron therapy in iron-deficient patients with systolic heart failure: a meta-analysis of randomized controlled trials. Eur J Heart Fail. 2016 Jul;18(7):786-95. doi: 10.1002/ejhf.473. Epub 2016 Jan 28. PMID 26821594
- [Background] Ponikowski P, Kirwan BA, Anker SD, Dorobantu M, Drozdz J, Fabien V, Filippatos G, Haboubi T, Keren A, Khintibidze I, Kragten H, Martinez FA, McDonagh T, Metra M, Milicic D, Nicolau JC, Ohlsson M, Parhomenko A, Pascual-Figal DA, Ruschitzka F, Sim D, Skouri H, van der Meer P, Jankowska EA. Rationale and design of the AFFIRM-AHF trial: a randomised, double-blind, placebo-controlled trial comparing the effect of intravenous ferric carboxymaltose on hospitalisations and mortality in iron-deficient patients admitted for acute heart failure. Eur J Heart Fail. 2019 Dec;21(12):1651-1658. doi: 10.1002/ejhf.1710. Epub 2019 Dec 28. PMID 31883356
- [Background] Ponikowski P, Kirwan BA, Anker SD, McDonagh T, Dorobantu M, Drozdz J, Fabien V, Filippatos G, Gohring UM, Keren A, Khintibidze I, Kragten H, Martinez FA, Metra M, Milicic D, Nicolau JC, Ohlsson M, Parkhomenko A, Pascual-Figal DA, Ruschitzka F, Sim D, Skouri H, van der Meer P, Lewis BS, Comin-Colet J, von Haehling S, Cohen-Solal A, Danchin N, Doehner W, Dargie HJ, Motro M, Butler J, Friede T, Jensen KH, Pocock S, Jankowska EA; AFFIRM-AHF investigators. Ferric carboxymaltose for iron deficiency at discharge after acute heart failure: a multicentre, double-blind, randomised, controlled trial. Lancet. 2020 Dec 12;396(10266):1895-1904. doi: 10.1016/S0140-6736(20)32339-4. Epub 2020 Nov 13. PMID 33197395
- [Background] Richards T, Baikady RR, Clevenger B, Butcher A, Abeysiri S, Chau M, Macdougall IC, Murphy G, Swinson R, Collier T, Van Dyck L, Browne J, Bradbury A, Dodd M, Evans R, Brealey D, Anker SD, Klein A. Preoperative intravenous iron to treat anaemia before major abdominal surgery (PREVENTT): a randomised, double-blind, controlled trial. Lancet. 2020 Oct 24;396(10259):1353-1361. doi: 10.1016/S0140-6736(20)31539-7. Epub 2020 Sep 5. PMID 32896294
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Durand E, Doutriaux M, Bettinger N, Tron C, Fauvel C, Bauer F, Dacher JN, Bouhzam N, Litzler PY, Cribier A, Eltchaninoff H. Incidence, Prognostic Impact, and Predictive Factors of Readmission for Heart Failure After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2017 Dec 11;10(23):2426-2436. doi: 10.1016/j.jcin.2017.09.010. PMID 29217006
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053